CLINICAL TRIAL: NCT03238612
Title: A Double-blind Randomised Controlled Trial on Flufenamic Acid for Hospitalised Influenza Infection
Brief Title: Flufenamic Acid for Hospitalised Influenza Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 16-418
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Influenza A
Keywords: influenza; FFA; clarithromycin; mortality; hospitalisation
MeSH Terms: conditions — Influenza, Human | interventions — Fatty Acids, Nonesterified; Clarithromycin; Oseltamivir; Antiviral Agents

STUDY DESIGN:
Intervention Model Description: Prospective Randomised Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFA, clarithromycin, oseltamivir (Experimental): oseltamivir 75mg + clarithromycin 500mg + FFA 200mg all twice daily for 2 days, followed by oseltamivir 75mg twice daily for 3 days
  Interventions: Drug: FFA, clarithromycin, oseltamivir
- Oseltamivir alone (Placebo Comparator): oseltamivir 75mg + two placebo capsules (identical in appearance to clarithromycin and FFA capsules respectively) twice daily for 2 days, followed by oseltamivir 75mg twice daily for 3 days
  Interventions: Drug: Oseltamivir alone

INTERVENTIONS:
Drug: FFA, clarithromycin, oseltamivir — 2-day course of triple combination of clarithromycin 500mg, flufenamic acid 200mg and oseltamivir 75mg twice daily followed by oseltamivir 75mg twice daily for 3 days
  Other Names: Antiviral combo
  Arms: FFA, clarithromycin, oseltamivir
Drug: Oseltamivir alone — 2-day course of oseltamivir 75mg plus placebo capsules twice daily followed by oseltamivir 75mg twice daily for 3 days as control
  Other Names: Antiviral
  Arms: Oseltamivir alone

SUMMARY:
It is well recognized that respiratory viruses cause substantial disease burden every year. Among all known respiratory viruses, influenza virus is the greatest cause of disability-adjusted life years lost, excess hospitalizations, and deaths in the elderly and patients with chronic illness. These patients are frequently hospitalized for pneumonia secondary to these respiratory viral infection. Recently, macrolide antimicrobial clarithromycin and flufenamic acid (FFA) have been shown to inhibit seasonal influenza virus infection in human airway epithelial cells with additional anti-inflammatory effect.

The investigators therefore plan to conduct a 3-year prospective study among adult patients hospitalized in Queen Mary Hospital for influenza with secondary pneumonia and randomized them to receive a course of oseltamivir + FFA + clarithromycin (as treatment) vs. a course of oseltamivir (current standard treatment as control). The objective of this prospective double-blind randomized controlled trial is to evaluate the efficacy of clarithromycin and FFA antiviral therapy in patients diagnosed to have pneumonia secondary to influenza infection.

DETAILED DESCRIPTION:
This double blind randomized-controlled trial will assess the clinical efficacy, mortality reduction and viral load reduction of clarithromycin and FFA in patients hospitalized for pneumonia secondary to influenza infection.

The investigators plan to enroll at least 200 adult patients. Enrolled patients will be randomized into 2 groups. Group 1: oseltamivir 75mg + clarithromycin 500mg + FFA 200mg all twice daily for 2 days, followed by oseltamivir 75mg twice daily for 3 days ; Group 2: oseltamivir 75mg + two placebo capsules (identical in appearance to clarithromycin and FFA capsules respectively) twice daily for 2 days, followed by oseltamivir 75mg twice daily for 3 days. The placebo capsules will contain inactive starch. All patients will receive a 5-day course of amoxicillin-clavulanate 1g bid for empirical coverage of community acquired pneumonia and esomeprazole 20mg daily for prevention of non-steroidal anti-inflammatory drugs related gastropathy.

Randomized treatment will be double blinded. Patients will be assigned to serial number by the study-coordinator. Each serial number will be linked to a computer-generated randomization list assigning the antiviral treatment regimens. The study medications will be dispensed by the hospital pharmacy and then to the patients by the medical ward nurses who will not know the treatment regimen of any subsequent patients. Enrolled patients could not differentiate the study or the placebo medication capsule which will be identical in appearance. The placebo capsules will contain inactive starch.

There will be 50% chance of random assignment into one of the treatment or control arms.

Clinical data, nasopharyngeal aspirate (NPA) and blood specimens will be collected daily if possible from admission till discharge, transfer to convalescent hospitals or death. All enrolled patients will be invited to the Infectious Disease outpatient clinic in Queen Mary Hospital for follow-up at 1 and 3 months after discharge. The investigators will retrieve your clinical information from the Clinical Medical System in the Queen Mary Hospital during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include all adult patients ≥18 years hospitalised for virologically confirmed influenza infection.
2. Auditory temperature ≥38°C with at least one of the following symptoms (cough, sputum production, sore-throat, nasal discharge, myalgia, headache or fatigue) upon admission
3. Symptom duration ≤72 hours
4. Radiological changes of pulmonary infiltrate by chest radiography or computerised tomography
5. All subjects give written informed consent. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterise immune response.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Allergy or severe reactions including renal or hepatic dysfunctions to clarithromycin, FFA, oseltamivir, amoxicillin-clavulanate or esomeprazole will be excluded
3. Patient with moderate renal impairment (creatinine clearance <30mL/min)
4. Prolonged QT or ventricular cardiac arrhythmias, including torsade de pointes.
5. Patient with a history of cholestatic jaundice and/or liver dysfunction associated with prior clarithromycin use
6. Patient on cisapride, pimozide, astemizole, terfenadine, ergotamine, dihyroergotamine, or statins medications which could not be stopped
7. Patient on colchicine with renal or hepatic impairment.
8. Pregnant or lactating women
9. Inability to comprehend and to follow all required study procedures
10. Have known human immunodeficiency virus infection
11. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.
12. Have a history of alcohol or drug abuse in the last 5 years. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days from commencement of treatment intervention
  30-day mortality

SECONDARY OUTCOMES:
NPA | 5 days post treatment
  nasopharyngeal aspirate viral load changes post treatment
PSI | 5 days post treatment
  Pneumonia severity index changes post treatment
Hospitalisation | Days of the subject hospitalised for the current admission up to 30 days
  Length of hospitalisation
AE | 2 weeks from subjects received treatment intervention
  Adverse events during treatment
Long-term mortality | 90 days from commencement of treatment intervention
  90-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- Ivan Hung, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hung IFN, To KKW, Chan JFW, Cheng VCC, Liu KSH, Tam A, Chan TC, Zhang AJ, Li P, Wong TL, Zhang R, Cheung MKS, Leung W, Lau JYN, Fok M, Chen H, Chan KH, Yuen KY. Efficacy of Clarithromycin-Naproxen-Oseltamivir Combination in the Treatment of Patients Hospitalized for Influenza A(H3N2) Infection: An Open-label Randomized, Controlled, Phase IIb/III Trial. Chest. 2017 May;151(5):1069-1080. doi: 10.1016/j.chest.2016.11.012. Epub 2016 Nov 22. PMID 27884765
- [Background] Hung IFN, To KKW, Lee CK, Lee KL, Yan WW, Chan K, Chan WM, Ngai CW, Law KI, Chow FL, Liu R, Lai KY, Lau CCY, Liu SH, Chan KH, Lin CK, Yuen KY. Hyperimmune IV immunoglobulin treatment: a multicenter double-blind randomized controlled trial for patients with severe 2009 influenza A(H1N1) infection. Chest. 2013 Aug;144(2):464-473. doi: 10.1378/chest.12-2907. PMID 23450336
- [Background] Li IW, Hung IF, To KK, Chan KH, Wong SS, Chan JF, Cheng VC, Tsang OT, Lai ST, Lau YL, Yuen KY. The natural viral load profile of patients with pandemic 2009 influenza A(H1N1) and the effect of oseltamivir treatment. Chest. 2010 Apr;137(4):759-68. doi: 10.1378/chest.09-3072. Epub 2010 Jan 8. PMID 20061398
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066